CLINICAL TRIAL: NCT00653705
Title: The Effect of Daily Consumption of Yogurt Containing Bifidobacterium Lactis (BB12) on Children's' Health and Child Care Absenteeism
Brief Title: The Effect of Yogurt Containing BB12 on Children's Health and Child Care Absenteeism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: General Mills (Industry)
Responsible Party: Principal Investigator, Tamar Ringel-Kulka, MPH, Assistant Professor, Maternal and Child Health, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 06-0901
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Last update posted 2013-05-31 (Estimated); Status verified 2013-05

CONDITIONS: Children's Health and Growth; Childcare Absenteeism
Keywords: Probiotics; Children; Child Care Center; Nutrition; Health promotion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Probiotic (Active Comparator): Children given probiotic BB12 enriched yogurt drink.
  Interventions: Other: Yogurt drink with probiotic bacteria BB12
- Control (Placebo Comparator): Children given dairy drink.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Yogurt drink with probiotic bacteria BB12 — Probiotic yogurt dairy drink with Bifidobacterium Lactis and prebiotics. One bottle a day for 16 weeks.
  Arms: Probiotic
Other: Placebo — Vanilla flavored dairy drink. One bottle a day for 16 weeks.
  Arms: Control

SUMMARY:
The aim of our study is to assess the effect of daily consumption of yogurt containing probiotic bacteria BB12 on the health and growth of healthy children 12-48 months of age in out of home child care.

ELIGIBILITY:
Inclusion Criteria:

* An informed consent has been signed by the parents.
* The child is at least one year old and has not had his 4th birthday at the beginning of the study
* The child is healthy.
* The child attends child care center at least 5 days a week, > 4 hours per day.

Exclusion Criteria:

* Was born preterm.
* Had a birth weight <2,500 g.
* Has congenital anomalies.
* Has a structural abnormality of the digestive tract or previous significant gastrointestinal surgery.
* Has chronic disease or malignancy.
* Has a serious, unstable medical condition.
* Is Failure to Thrive (FTT) (<5th percentile of ideal body weight).
* Has an allergy or atopic disease.
* Has an allergy or intolerance to milk/dairy products.
* Has an established diagnosis of lactase deficiency.
* Is predisposed to infection (i.e., compromised immune system, HIV-AIDS, active bacterial disease, under steroid treatment).
* Received antibiotic treatment or intentionally consumes probiotic products during the preceding 4 weeks. (If the subject was on antibiotics before the beginning of the study or probiotics, a washout period of 2 weeks is required.)

Ages: 12 Months to 48 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 181 (Actual)
Dates: Start 2007-01; Primary Completion 2008-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Days of illness symptoms, number, duration and severity of illness episodes, day care absenteeism, and parental work absenteeism | 16 weeks

SECONDARY OUTCOMES:
Health care utilization and illness related costs as measured by number of physician visits, ER visits, hospitalizations, and antibiotics use. Also, child growth and quality of life. Exploratory biomarker outcomes in stool. | 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Tamar Ringel-Kulka, MD, MPH, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, School of Public Health, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Ringel-Kulka T, Kotch JB, Jensen ET, Savage E, Weber DJ. Randomized, double-blind, placebo-controlled study of synbiotic yogurt effect on the health of children. J Pediatr. 2015 Jun;166(6):1475-81.e1-3. doi: 10.1016/j.jpeds.2015.02.038. Epub 2015 Apr 1. PMID 25841539